CLINICAL TRIAL: NCT06554132
Title: Investigation of Respiratory Muscle Strength and Aerobic Capacity in Patients With Scleroderma
Brief Title: Respiratory Muscle Strength and Aerobic Capacity in Scleroderma
Status: Recruiting | Type: Observational
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Firat University, Firat University
Other Study IDs: 2024/10-02
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Scleroderma
Keywords: Scleroderma; Respiratory muscle strength; Aerobic capacity
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scleroderma group: Scleroderma patients will be evaluated in terms of respiratory muscle strength, aerobic capacity, pulmonary function test and fatigue.
  Interventions: Other: Scleroderma Group
- Healthy group: Healthy people will be evaluated in terms of respiratory muscle strength, aerobic capacity, pulmonary function test and fatigue.
  Interventions: Other: Healthy group

INTERVENTIONS:
Other: Scleroderma Group — Scleroderma patients will be evaluated in terms of respiratory muscle strength, aerobic capacity, pulmonary function test and fatigue.
  Groups: Scleroderma group
Other: Healthy group — Healthy people will be evaluated in terms of respiratory muscle strength, aerobic capacity, pulmonary function test and fatigue.
  Groups: Healthy group

SUMMARY:
Primary aim of this study was to compare respiratory muscle strength, aerobic capacity, dyspnea, pulmonary function tests and fatigue values with healthy controls. The secondary aim was to evaluate the relationship between respiratory muscle strength and other parameters in these patients and to examine the factors that may affect respiratory muscle strength. Respiratory muscle strength, aerobic capacity, respiratory function tests and fatigue will be evaluated

DETAILED DESCRIPTION:
Scleroderma is a systemic connective tissue disease characterized by progressive thickening of the skin, the etiology of which has not been fully elucidated, in which microvascular damage, immune activation and fibrosis play a role. Primary aim of this study was to compare respiratory muscle strength, aerobic capacity, dyspnea, pulmonary function tests and fatigue values with healthy controls. The secondary aim was to evaluate the relationship between respiratory muscle strength and other parameters in these patients and to examine the factors that may affect respiratory muscle strength. The study will include 15 patients and 15 healthy individuals of the same age and gender. Respiratory muscle strength, aerobic capacity, respiratory function tests and fatigue will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Ssk according to ACR/EULAR criteria
* Stable medical treatment for 3 months

Exclusion Criteria:

* Having a regular exercise habit (doing regular exercise at least once a week for the last 3 months)
* Comorbidity with another chronic disease that may affect aerobic capacity or respiratory muscle strength
* Having concomitant acute respiratory diseases
* Having a smoking habit
* History of orthopedic or neurologic disease in the lower extremities that may prevent cycling

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who have not a chronic disease or othopedic disease will be included as Healthy controls
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength assessment | 5 minutes
  Respiratory muscle strength will be assessed with an intraoral pressure gauge. These are the intraoral pressures measured at maximal respiration against a valve that closes the airways. When applying MIP, the patient is asked to perform maximal expiration. As a result, the patient is asked to maximally inspire against the closed airway and maintain this for 1-3 seconds. MEP, on the other hand, after maximal inspiration, the patient is asked to perform maximal expiration against the closed airway for 1-3 seconds.

SECONDARY OUTCOMES:
Aerobic capacity assessment | 10 minutes
  Aerobic capacity will be assessed using exercise testing. VO2max will be assessed using the Cosmed FitMate Pro® (Cosmed, Italy). The FitMate Pro® includes a turbine flowmeter to measure ventilation and a galvanic fuel cell oxygen sensor to analyze the oxygen fraction in expired gases.
Fatigue assessment | 2 minutes
  Fatigue will be assessed with the Fatigue Severity Scale (FSS), the Turkish validity and reliability of which was performed by Armutlu et al. This scale includes 9 questions related to fatigue.
Pulmonary function test | 5 minutes
  Pulmonary function test is routinely performed in Ssk patients. FEV1, DLCO and FEV1/FVC values will be recorded from the patients' files.

CONTACTS AND LOCATIONS:
Locations (1):
- Songul Baglan Yentur, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No